# ADDENDUM TO STATISTICAL ANALYSIS PLAN

#### Clinical Trial

A multicenter, multinational, randomized, controlled, assessor blinded study, performed in subjects with thermal burns, to evaluate the efficacy and safety of NexoBrid compared to Gel Vehicle and compared to Standard of Care (DETECT)

Sponsor:

MediWound, Ltd.

42 Hayarkon Street

North Industrial Area

Yavne, Israel 8122745

Trial protocol code: MW2010-03-02

EudraCT number: 2014-001672-55

IND No.: 65,448



Competence Center for Clinical Trials Bremen - Biometry

Author: Dr. Martin Scharpenberg

Version of 26 February 2020, Addendum to Version V03

# 1. Table of Contents

| 1. | . Tabl | Table of Contents | |
|----|----------|----------------------------|---|
| 2. | Stud | y Administrative Structure | 3 |
| | 2.1. | Sponsor | 3 |
| | 2.2. | Study Conduct | 3 |
| | 2.3. | Statistics | 4 |
| 3. | . Sign | atures | 5 |
| 4. | . List o | of Abbreviations | 6 |
| 5. | . Ratio | onale for the Addendum | 7 |

## 2. Study Administrative Structure

## 2.1. Sponsor

Sponsor: MediWound, Ltd

42 Hayarkon Street North Industrial Area Yavne, Israel 8122745

Represented by: Prof. Lior Rosenberg

**Chief Medical Officer** 

MediWound Ltd.

Keren David Zarbiv

**Director Clinical Affairs** 

MediWound Ltd.

Nimrod Leuw

Director of QA/QC MediWound Ltd.

## 2.2. Study Conduct

Study Conduct (CRO): Dr. Marco Schwarzer

GCP-Service International Ltd. & Co. KG

Anne-Conway-Str. 2

28359 Bremen

## 2.3. Statistics

Statisticians: Prof. Dr. h.c. Jürgen Timm

Dr. Martin Scharpenberg

Competence Center for Clinical Trials Bremen

University of Bremen

Linzer Str. 4

28359 Bremen

Germany

## 3. Signatures

Keren David Zarbiv

Sponsor Representative MediWound Ltd.

Keren David

02.03.2020

Date

Dr. Marco Schwarzer

Study Conduct (CRO) GCP-Service International Ltd. & Co. KG Luan

Signature

Signature

Prof. Dr. h.c. Jürgen Timm

Principal Statistician

Competence Center for Clinical Trials Bremen, University of Bremen

Signature

Date

Dr. Martin Scharpenberg

Statistician/Author

Competence Center for Clinical Trials Bremen, University of Bremen

# 4. List of Abbreviations

| abbreviation | meaning |
|--------------|----------------------------------------------|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| BLA | Biologics License Application |
| CSR | Clinical Study Report |
| FDA | Food and Drug Administration |
| INR | International Normalized Ratio |
| ITT | Intention to Treat |
| KKSB | Competence Center for Clinical Trials Bremen |
| PT | Preferred Term |
| PTT | Prothrombin Time |
| SAE | Serious Adverse Event |
| SOC | System Organ Class |
| TEAE | Treatment Emergent Adverse Event |
| TESAE | Treatment Emergent Serious Adverse Event |
| TW | Target Wound |

#### 5. Rationale for the Addendum

This addendum describes safety data analyses to be performed in addition to the final SAP (Version 3, 29 November 2018). The decision to add these analyses was made after breaking the blinding and in knowledge of the primary statistical analysis results computed in accordance with the SAP.

All originally planned analyses, as described in the final SAP, version 3, were performed and summarized in a Statistical Analysis Report dated 20 June 2019. Changed outputs described in this document will be implemented in the study CSR. The sponsor requested these ad hoc analyses in order to support the interpretation of the safety data statistical analysis results and to fulfil the FDA request for treatment emergent Adverse Events analysis as noted in the pre-BLA meeting minutes.

Furthermore, the calculation of some variables is adapted to be conform with the Analysis Data Model (ADaM) Implementation Guide v1.1. and to be consistent throughout the analysis.

## 6. General changes

Some general changes to the layout of tables described in the SAP will be performed:

- For some tables, the treatment arms will be presented in columns rather than rows, to facilitate between-treatment-group comparisons.
- Descriptive statistics tables will be combined for some baseline characteristics.
- The number of censored observation will be added to the tables of descriptive statistics for time to event endpoints.

Statistical analyses for all safety parameters which were described in the SAP are included in the Statistical analysis report, yet will not be included in appendix 14 of the CSR and is available upon request.

Furthermore, the calculation of some variables is adapted as follows to be conform with the Analysis Data Model (ADaM) Implementation Guide v1.1. and to be consistent throughout the study:

- AGE (Age) = RFICDTC (Date of Informed Consent) BRTHDTC (Date of Birth)
   In the SAP, the date of physical examination instead of the date of informed consent is used which leads to missing age for two screening failures.
- CHG (Change from baseline) = AVAL (Analysis Value) BASE (Baseline Value)

According to the SAP, the change from baseline should be calculated as BASE – AVAL which is not conform with the ADaM Implementation Guide. The calculation of pre-post differences is adapted accordingly (i.e. pre-post difference = post value – pre-value) to be consistent with the calculation of the change from baseline. However, the calculation described in the SAP will still be done (variable: BCHG) and form the basis of the analyses presented in the CSR.

## 7. Additional Analyses

## 7.1. Central Laboratory values

Shift tables for central laboratory values indicating shifts from baseline to post every type of eschar removal procedure (first application, additional application, surgical application, additional surgical application, and nonsurgical application) will be produced (see Table 1).

Furthermore, shift tables indicating shifts from baseline to any low/high or no low/high values will be presented (see Table 2).

Additional tables will indicate shifts from baseline to any post treatment clinically significant result (see Table 3). A listing of subjects experiencing such shifts will be provided.

The above tables will be presented for biochemistry parameters, hematology parameters and urine analysis parameters separately, and for parameters with numeric values only.

## 7.2. Local Laboratory values

The following sets of tables will be produced separately for INR and PTT:

- Shift tables indicating shifts from baseline to post first application, 24 hours past start and 48 hours past start, similar to Table 1
- Shift tables indicating shifts from baseline to any low/high or no low/high values post treatment (see Table 2) as well as a listing of subject experiencing such shifts
- Shift tables indicating shifts from baseline to any post treatment clinically significant result (see Table 3) as well as a listing of subjects experiencing such shifts

## 7.3. Vital signs

For the vital signs assessments, shift tables will be produced indicating shifts from baseline to any post-treatment time point (post first treatment, post second treatment, and post third treatment), as well as to the daily assessments for day 1 to day 7 (see Table 4).

Furthermore, shift tables indicating shifts from baseline to any post treatment clinically significant result (as in Table 3) will be provided. A subject listing of patients experiencing such shifts will be provided.

#### 7.4. Pain

For the pain assessment, shift tables will be produced indicating the shift from baseline to pre and post any treatment time point (first application, additional application, surgical application, additional surgical application, and nonsurgical application), as well as to the daily assessments for day 1 to day 7 (see Table 4).

Furthermore, shift tables indicating shifts from baseline to any post treatment clinically significant result (see Table 5) will be provided.

#### 7.5. Adverse Events

The following tables will be produced in addition to the tables described in the SAP:

- Summary of Treatment Emergent Adverse Events (TEAEs) on a subject level (see Table 6)
- Summary of TEAEs by System Organ Class (SOC), and Preferred Term (PT) (see Table 7) separately for:
  - All TEAEs
  - Treatment related TEAEs
  - General TEAEs
  - Local, not TW-related TEAEs
  - Local, TW-related TEAEs
  - TEAEs with PTs related to fever (Pyrexia, Body Temperature Increased, Hypothermia)
  - TEAEs with Target Wound Infections (only if Local, TW-related: Wound Infection Bacterial, Staphylococcal Skin Infection, Wound Infection, Wound Infection Staphylococcal)
  - Pain TEAEs (Pain: Pain; Post-traumatic pain; Uncontrolled pain in TW1,2 and
     3; Pain in extremity [if Local, TW-related])

- o TEAEs including Tachycardia PTs (Sinus Tachycardia, Tachycardia)
- Summary of TEAEs by SOC, PT, and time of onset (see Table 8) separately for:
  - o All TEAEs
  - General TEAEs
  - o Local, not TW-related TEAEs
  - Local, TW-related TEAEs
  - All Treatment Emergent Serious Adverse Events (TESAEs)
- Summary of TEAE by SOC, PT and maximum intensity (see Table 9). In this table, patients who experienced multiple AEs with the same PT, but different intensities will be counted only once per PT with their maximum intensity. Subjects with multiple AEs with the same SOC but different intensities will be counted only once per SOC with their maximum intensity in the SOC row. This table will be produced separately for:
  - o All TEAEs
  - Treatment related TEAEs
  - General Treatment related TEAEs
  - Local, not TW-related Treatment related TEAEs
  - Local, TW-related Treatment related TEAEs
  - All TESAEs
  - Treatment related TESAEs

All AE/SAE/TEAE/TESAE tables will be produced separately for Adverse Events occurring in the acute phase, in the second stage (3-12 months), and combined for the time frame 0-12 months.

## 7.6. Subgroup Analysis

## 7.6.1. Target wounds in the anatomical area of the hand

Additional to the subgroup analysis described in the SAP, which was defined on a subset of target wounds, the primary and secondary endpoint were also analyzed on a patient level using the subgroup of patients having at least one target wound that is found, at least partly, in the anatomical area of the hand.

## 7.6.1. Target wounds that are entirely full thickness

Additional to the subgroup analysis described in the SAP, which was defined on a subset of target wounds (i.e. all target wounds that are entirely full thickness), the primary and secondary endpoint were also analyzed on a patient level using the subgroup of patients having at least one target wound that is entirely full thickness.

# 8. Lay-out and list of tables

Table 1: Laboratory Value Shift Table for Changes from Baseline

| | | | | | Time poi | int | |
|---|---|---|---|---|---|---|---|
| Lab Value | Treatment | Baseline | Low:<br><32<br>n (%) | Normal:<br>32-50<br>n (%) | High:<br>>50<br>n (%) | Missing<br>n (%) | Total<br>n (%) |
| √alue [unit] | NexoBrid<br>(N = xxx) | <32 | | | | | |
| | | 32-50 | | | | | |
| | | >50 | | | | | |
| | | Missing | | | | | |
| | | Total | | | | | |
| /alue [unit] | SOC<br>(N = xxx) | <32 | | | | | |
| | | 32-50 | | | | | |
| | | >50 | | | | | |
| | | Missing | | | | | |
| | | Total | | | | | |

| | | | | | Time po | int | |
|---|---|---|---|---|---|---|---|
| Lab Value | Treatment | Baseline | Low:<br><32<br>n (%) | Normal:<br>32-50<br>n (%) | High:<br>>50<br>n (%) | Missing<br>n (%) | Total<br>n (%) |
| Value [unit] | Gel Vehicle<br>(N = xxx) | <32 | | | | | |
| | | 32-50 | | | | | |
| | | >50 | | | | | |
| | | Missing | | | | | |
| | | Total | | | | | |

N = number of subjects with the respective eschar removal procedure; N/A = not applicable, n = number of subjects with respective category, % = n/N\*100

Program: xxx.sas / Output run time: xxx / Data Base Extraction Date xxx

Output File: xxx.rtf

Table 2: Laboratory Value Shift Table, Shift to Any Low or High

| | | | Any post-treatment time point | | | |
|---|---|---|---|---|---|---|
| Lab Value | Treatment | Baseline | Any Low<br>n (%) | No Low<br>n (%) | Any High<br>n (%) | No High<br>n (%) |
| /alue [unit] | NexoBrid<br>(N = xxx) | Low | | | | |
| | | Normal | | | | |
| | | High | | | | |
| | | Missing/not applicable | | | | |
| | | Total | | | | |
| Value [unit] | SOC<br>(N = xxx) | Low | | | | |
| | | Normal | | | | |
| | | High | | | | |
| | | Missing/not applicable | | | | |
| | | Total | | | | |
| Value [unit] | Gel Vehicle<br>(N = xxx) | Low | | | | |
| | | Normal | | | | |

| | | | Any post-treatment time point | | | |
|---|---|---|---|---|---|---|
| Lab Value | Treatment | Baseline | Any Low<br>n (%) | No Low<br>n (%) | Any High<br>n (%) | No High<br>n (%) |
| | | High | | | | |
| | | Missing/not applicable | | | | |
| | | Total | | | | |

N = number of subjects with the respective eschar removal procedure, n = number of subjects with respective category, % = n/N\*100

Program: xxx.sas / Output run time: xxx / Data Base Extraction Date xxx

Output File: xxx.rtf

Table 3: Laboratory Value Shifts from Baseline to Any Post-treatment Clinically Significant Result

| | | | | Any post-treat | ment time po | oint |
|---|---|---|---|---|---|---|
| Lab Value | Treatment | Baseline | Any pCS<br>low<br>n (%) | No pCS low<br>n (%) | Any pCS<br>high<br>n (%) | No pCS<br>high<br>n (%) |
| pCS low:<br>pCS high: | | | | | | |
| Value [unit] | NexoBrid<br>(N = xxx) | Low | | | | |
| | | Normal | | | | |
| | | High | | | | |
| | | Missing/not applicable | | | | |
| | | Total | | | | |
| Value [unit] | SOC<br>(N = xxx) | Low | | | | |
| | | Normal | | | | |
| | | High | | | | |
| | | Missing/not applicable | | | | |
| | | Total | | | | |
| Value [unit] | Gel Vehicle<br>(N = xxx) | Low | | | | |

Normal

High

Missing/not applicable

Total

N = number of subjects in the Safety Population, n = number of subjects with respective category, % = n/N\*100 N/A = not applicable; ULN = upper limit of normal pCS = potentially Clinically Significant

Program: xxx.sas / Output run time: xxx / Data Base Extraction Date xxx

Output File: xxx.rtf

Table 4: Vital Sings/Pain Changes from Baseline by Time Point

| | | | | | | E | Baseline A | ssessme | ents | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | NexoBrid (N= XXX) | | Standard of Care (N= XXX) | | | Gel (N= XXX) | | | | | |
| Time<br>point | Assessment | <90<br>n (%) | 90-180<br>n (%) | >180<br>n (%) | Missin<br>g<br>n (%) | <90<br>n (%) | 90-180<br>n (%) | >180<br>n (%) | Missin<br>g<br>n (%) | <90<br>n (%) | 90-180<br>n (%) | >180<br>n (%) | Missin<br>g<br>n (%) |

Post first pCS (Low) treatment

no pCS

pCS (High)

Missing

Total

N = number of subjects in the Safety Population, n = number of subjects with respective category, % = n/N\*100 pCS = potentially Clinically Significant

Program: xxx.sas / Output run time: xxx / Data Base Extraction Date xxx

Output File: xxx.rtf

Table 5: Pain Assessment Clinically Significant Results Shifts from Baseline to Any Post-treatment Time Point

| | | | A | ny post-treat | ment time po | int |
|---|---|---|---|---|---|---|
| Visual Analog Scale | Treatment | Baseline | Any<br>abnormal<br>(nCS)<br>n (%) | No<br>abnormal<br>(nCS)<br>n (%) | Any<br>abnormal<br>(CS)<br>n (%) | No<br>abnormal<br>(CS)<br>n (%) |
| Dain Interesity (see | Nava Deid | A la a a l | | | | |
| Pain Intensity (mm) | NexoBrid<br>(N = XXX) | Abnormal<br>(nCS) | | | | |
| | | Normal | | | | |
| | | Abnormal<br>(CS) | | | | |
| | | Missing/not applicable | | | | |
| | | Total | | | | |
| Pain Intensity (mm) | SOC<br>(N = XXX) | Abnormal<br>(nCS) | | | | |
| | | Normal | | | | |
| | | Abnormal<br>(CS) | | | | |
| | | Missing/not applicable | | | | |
| | | Total | | | | |

| | | | A | ny post-treat | ment time po | oint |
|---|---|---|---|---|---|---|
| Visual Analog Scale | Treatment | Baseline | Any<br>abnormal<br>(nCS)<br>n (%) | No<br>abnormal<br>(nCS)<br>n (%) | Any<br>abnormal<br>(CS)<br>n (%) | No<br>abnormal<br>(CS)<br>n (%) |
| Pain Intensity (mm) | Gel Vehicle<br>(N = XXX) | Abnormal<br>(nCS) | | | | |
| | | Normal | | | | |
| | | Abnormal<br>(CS) | | | | |
| | | Missing/not applicable | | | | |
| | | Total | | | | |

N = number of subjects in the Safety Population, n = number of subjects with respective category, % = n/N\*100

Program: xxx.sas / Output run time: xxx / Data Base Extraction Date xxx

Output File: xxx.rtf

## Table 6: Summary of Treatment Emergent Adverse Events - Patient level

| Treatment | | | | | |
|---|---|---|---|---|---|
| | NexoBrid<br>=XXX) | of C | dard<br>Care<br>XXX) | Topica<br>Veh<br>(N=X | icle |
| n | % | n | % | n | % |

With at least one TEAE

With at least one mild or moderate TEAE

With at least one severe TEAE

With at least one TESAE

With at least one TEAE not related or remotely related to study drug

With at least one TEAE possibly, probably, or related to study drug

With treatment-emergent outcome of death

N = number of subjects in the Safety Population, n = number of subjects with respective category, % = n/N\*100

Program: xxx.sas / Output run time: xxx / Data Base Extraction Date xxx

Output File: xxx.rtf

Table 7: Summary of TEAEs/TESAEs by System Organ Class and Preferred Term

| System Organ Class<br>Preferred Term | Topical:NexoBrid<br>Gel (N=XXX)<br>n (%) | Standard<br>of Care<br>(N=XXX)<br>n (%) | Topical:Gel<br>Vehicle<br>(N=XXX)<br>n (%) |
|---|---|---|---|
|---|---|---|---|

System Organ Class 1

Preferred Term 1

Preferred Term 2

Preferred Term 3

Preferred Term 4

System Organ Class 2

Preferred Term 1

Preferred Term 2

N = number of subjects in the Safety Population, n = number of subjects with respective category, % = n/N\*100

Program: xxx.sas / Output run time: xxx / Data Base Extraction Date xxx

Output File: xxx.rtf

Table 8: Summary of TEAEs/TESAEs by System Organ Class, Preferred Term and Time of Onset

| System Organ Class<br>Preferred Term | Time of Onset | Topical:NexoBrid Gel<br>(N=xxx)<br>n (%) | Standard of<br>Care (N=xxx)<br>n (%) | Topical:Gel<br>Vehicle (N=xxx<br>n (%) |
|---|---|---|---|---|
| System Organ Class 1 | Total | | | |
| | During the treatment session | | | |
| | 1st week after treatment | | | |
| | Week 2 - 4 after treatment | | | |
| | Week 5 - 8 after treatment | | | |
| | Later | | | |
| | Missing | | | |
| Preferred Term 1 | Total | | | |
| | During the treatment session | | | |
| | 1st week after treatment | | | |
| | Week 2 - 4 after treatment | | | |
| | Week 5 - 8 after treatment | | | |
| | Later | | | |
| | Missing | | | |
| Preferred Term 2 | Total | | | |
| | During the treatment session | | | |

| System Organ Class<br>Preferred Term | Time of Onset | Topical:NexoBrid Gel<br>(N=xxx)<br>n (%) | Standard of<br>Care (N=xxx)<br>n (%) | Topical:Gel<br>Vehicle (N=xxx)<br>n (%) |
|---|---|---|---|---|
| | 1st week after treatment | | | _ |
| | Week 2 - 4 after treatment | | | |
| | Week 5 - 8 after treatment | | | |
| | Later | | | |
| | Missing | | | |

Adverse events are presented in alphabetic order of system organ class and descending order of preferred term in the Total row of the NexoBrid group

Classifications of Adverse Events are based on the MedDRA (version 21.1)

Program: xxx.sas / Output run time: xxx / Data Base Extraction Date xxx

Output File: xxx.rtf

Table 9: Summary of TEAEs/TESAEs by System Organ Class, Preferred Term and Maximum Intensity

| System Organ Class<br>Preferred Term | Topical:NexoBrid Gel (N=XXX)<br>n (%) | | | Standard of Care (N=XXX)<br>n (%) | | | Topical:Gel Vehicle (N=XXX)<br>n (%) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Mild | Moderate | Severe | Total | Mild | Moderate | Severe | Total | Mild | Moderate | Severe | Total |
| System Organ Class 1 | | | | | | | | | | | | |
| Preferred Term 1 | | | | | | | | | | | | |
| Preferred Term 2 | | | | | | | | | | | | |
| System Organ Class 2 | | | | | | | | | | | | |
| Preferred Term 1 | | | | | | | | | | | | |

AE is defined as related if causality is possibly related, probably related or related

Subjects are counted at the maximum severity level, only once in each system organ class category, and only once in each preferred term category Events are counted for maximum severity level on a patient level. If an event was reported multiple times in the same patient, only the maximum severity is counted.

Adverse events are presented in alphabetic order of system organ class and descending order of preferred term in the Total column of the NexoBrid group Classifications of Adverse Events are based on the MedDRA (version 21.1)

N = number of subjects in the Safety Population, n = number of subjects with respective category, % = n/N\*100

Program: xxx.sas / Output run time: xxx / Data Base Extraction Date xxx

Output File: xxx.rtf